CLINICAL TRIAL: NCT00528359
Title: Phase 1 Study of Insulin Sensitivity, Adjusted β-Cell Function and Adiponectin Among Lean Drug-naïve Schizophrenic Subjects Treated With Atypical Antipsychotic Drugs
Brief Title: β-Cell Function in Schizophrenic Subjects on Atypical Antipsychotic drugS
Acronym: SANAT
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Other Study IDs: AAD-001
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Schizophrenia
Keywords: antipsychotic drugs; schizophrenia; β-cell function; insulin resistance
MeSH Terms: conditions — Schizophrenia; Insulin Resistance | interventions — Quetiapine Fumarate; Olanzapine; Risperidone; Aripiprazole

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: 36 lean schizophrenic subjects free of metabolic syndrome(M:F 24:12; Caucasian n=23; North-African n=12; South-Asian n=1)aged 35±9 years
  Interventions: Drug: quetiapine or olanzapine or risperidone or aripiprazole

INTERVENTIONS:
Drug: quetiapine or olanzapine or risperidone or aripiprazole

SUMMARY:
The purpose of this study is to determine whether atypical antipsychotic drugs (commonly prescribed for treating schizophrenia) induce changes in anthropometry and metabolism, including alteration in insulin sensitivity and/or insulin secretion by the pancreas, when given to lean, non-diabetic, individuals who are antipsychotic drug(s)-naïve, and free of metabolic syndrome at enrollment.

DETAILED DESCRIPTION:
Atypical antipsychotic drugs (AADs) induce weight gain, truncal adiposity and may engender a metabolic syndrome which may progress to IFG/IGT or DM. AADs effects in lean schizophrenic patients without metabolic syndrome are not documented, especially the relationship between weight gain and changes in insulin sensitivity (S), beta-cell function (β), and circulating adiponectin. We prospectively determined the outcome of 9-month therapy with AADs on anthropometrics, metabolism and adiponectin, including HOMA-modeling of S, β, and βxS (hyperbolic product, assessing individual β adjusted for S)in 36 schizophrenic subjects (M:F 24:12; Caucasian n=23; North-African n=12; South-Asian n=1) aged 35±9 years (mean±1SD) free of MetS (NCEP-ATPIII).

ELIGIBILITY:
Inclusion Criteria:

* age 18-55 years
* body mass index <25.0 kg/m²
* waist circumference <102 (men) and <88 cm (women)
* absence of a metabolic syndrome according to NCEP ATPIII criteria
* normoglycaemic (fasting plasma glucose levels <100 mg/dl)

Exclusion Criteria:

* previous use of antipsychotic drugs
* concomitant therapy with drugs known to possess an inherent potential to increase weight and/or to alter glucose metabolism (including antihistaminic drugs, glucocorticoids, β-blockers, antiepileptic drugs and mirtazapine)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-10; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe M ORIOT, MD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Sanatia Hospital, Brussels, Belgium